CLINICAL TRIAL: NCT03754868
Title: Analysis of the Activity of Different Coagulation Factors and Monitoring of Coagulation Using Point-of-care Devices During a Veno-venous ECMO Therapy
Brief Title: Evaluation of Coagulation Factors and Point-of-care Devices During Veno-venous ECMO Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital Goettingen (Other)
Responsible Party: Principal Investigator, Saskia Wand, Resident for Anesthesiology, Principal Investigator, University Hospital Goettingen
Other Study IDs: 19/5/13
Record Dates: First submitted 2018-11-07; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Coagulation Factor Deficiency
Keywords: ECMO; Coagulation monitoring; point-of-care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detailed coagulation monitoring — Monitoring of coagulation using activity of coagulation factors, rotational thrombelastometry and multiple electrode aggregometry

SUMMARY:
Hemorrhagic and thromboembolic complications are common in Veno-venous ECMO therapy. The aim of this study is to provide a detailed analysis of the activity of different coagulation factors and changes in functional coagulation measurements as in rotational thrombelastometry and multiple electrode aggregometry in the course of ECMO therapy.

ELIGIBILITY:
Inclusion Criteria:

* Need for a Veno-venous extracorporeal membrane oxygenation therapy

Exclusion Criteria:

* Known coagulation disorders
* Refusal to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the need for Veno-venous ECMO therapy treated in a tertiary intensive care unit.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in the activity of coagulation factor II [%] during Veno-venous ECMO therapy | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor II in % through standard coagulometric methods.
Changes in the activity of coagulation factor V [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor V in % through standard coagulometric methods.
Changes in the activity of coagulation factor VII [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor VII in % through standard coagulometric methods.
Changes in the activity of coagulation factor VIII [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor VIII in % through standard coagulometric methods.
Changes in the activity of coagulation factor IX [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor IX in % through standard coagulometric methods.
Changes in the activity of coagulation factor X [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor X in % through standard coagulometric methods.
Changes in the activity of coagulation factor XII [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor XII in % through standard coagulometric methods.
Changes in the activity of coagulation factor XIII [%] during Veno-venous ECMO | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessment of the activity of coagulation factor XIII in % through standard coagulometric methods.

SECONDARY OUTCOMES:
vWF-Antigen | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Measurement of the vWF-Antigen
Changes in the vWF:Ristocetin-Cofaktor-Activity in % during Veno-venous ECMO therapy | Pre-canulation and 6 hours, 1 day, 3 days, 7 days, 11 days, 15 days and 21 days after canulation
  Repeated assessments of the vWF:Ristocetin-Cofaktor-Activity [%]
Changes in CT-EXTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clotting time (CT) in the extrinsically activated assay (EXTEM) of rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in CT-INTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clotting time (CT) in the intrinsically activated assay (INTEM) of rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in CT-FIBTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clotting time (CT) in the extrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of Cytochalasin D to inhibit platelet aggregation (FIBTEM), results were noted in seconds.
Changes in CT-HEPTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clotting time (CT) in the intrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of heparin to eliminate heparin effects (HEPTEM), results were noted in seconds.
Changes in CFT-EXTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clot formation time (CFT) in the extrinsically activated assay (EXTEM) of rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in CFT-INTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clot formation time (CFT) in the intrinsically activated assay (INTEM) of rotational thrombelastometry (ROTEM), results were noted in seconds.
Changes in CFT-FIBTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clot formation time (CFT) in the extrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of Cytochalasin D to inhibit platelet aggregation (FIBTEM), results were noted in seconds.
Changes in CFT-HEPTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in clot formation time (CFT) in the intrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of heparin to eliminate heparin effects (HEPTEM), results were noted in seconds.
Changes in MCF-EXTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in maximum clot firmness (MCF) in the extrinsically activated assay (EXTEM) of rotational thrombelastometry (ROTEM), results were noted in millimeters.
Changes in MCF-INTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in maximum clot firmness (MCF) in the intrinsically activated assay (INTEM) of rotational thrombelastometry (ROTEM), results were noted in millimeters.
Changes in MCF-FIBTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in maximum clot firmness (MCF) in the extrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of Cytochalasin D to inhibit platelet aggregation (FIBTEM), results were noted in millimeters.
Changes in MCF-HEPTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in maximum clot firmness (MCF) in the intrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of heparin to eliminate heparin effects (HEPTEM), results were noted in millimeters.
Changes in Alpha angle-EXTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in Alpha angle in the extrinsically activated assay (EXTEM) of rotational thrombelastometry (ROTEM), results were noted in degree.
Changes in Alpha angle-INTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in Alpha angle in the intrinsically activated assay (INTEM) of rotational thrombelastometry (ROTEM), results were noted in degree.
Changes in Alpha angle-FIBTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in Alpha angle in the extrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of Cytochalasin D to inhibit platelet aggregation (FIBTEM), results were noted in degree.
Changes in Alpha angle-HEPTEM | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Changes in Alpha angle in the intrinsically activated assay of rotational thrombelastometry (ROTEM) with the addition of heparin to eliminate heparin effects (HEPTEM), results were noted in degree.
Changes in arachidonic acid induced platelet aggregation assessed by multiple elcetrode aggregometry (MEA)(ASPItest) | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Platelet aggregation after stimulation with arachidonic acid was recorded in aggregational units (AU).
Changes in adenosine diphosphate (ADP) induced platelet aggregation assessed by multiple elcetrode aggregometry (MEA)(ADPtest) | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Platelet aggregation after stimulation with ADP was recorded in aggregational units (AU).
Changes in thrombin-receptor activating peptide (TRAP) induced platelet aggregation assessed by multiple elcetrode aggregometry (MEA)(TRAPtest) | Pre-canulation, 6 hours, 1 day, 2 days, 4 days, 7 days and 11 days after canulation
  Platelet aggregation after stimulation with TRAP was recorded in aggregational units (AU).
Light transmission aggregometry | 6 hours and 7 days after canulation
  Measurement of platelet function
Quick | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of Quick in %
activated partial thromboplastin time (aPTT) | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of aPTT in seconds
Fibrinogen | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of fibrinogen concentration in mg/dl
Platelet count | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of platelet count/µl
activated clotting time (ACT) | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of ACT in seconds
Antithrombin III (ATIII) | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  Measurement of ATIII in %
Measurement of Anti-Xa-Activity in % | Pre-canulation, 6 hours, 1 day, 2 days, 3 days, 4 days, 5, days, 6 days, 7 days, 10, days, 11 days 14 days, 17 days, 19 days and 21 days after canulation
  Measurement of Anti-Xa-Activity by chromogenic assay to determine heparin effect
D-Dimers | Pre-canulation, 6 hours, 1 day, 2 days, 3 days, 4 days, 5, days, 6 days, 7 days, 10, days, 11 days 14 days, 17 days, 19 days and 21 days after canulation
  Measurement of D-Dimers
hemoglobin | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  hemoglobin concentration in g/dl
leucocyte count | Pre-canulation, 6 hours and daily from day 1- day 21after canulation
  leucocyte count/µl
Hemorrhagic complications | Daily from day 1-21
  Structured documentation of hemorrhagic complications
Thrombotic complications | Daily from day 1-21
  Structured documentation of thrombotic complications
Oxygenator State | Daily from day 1-21
  Structured documentation of the state of the oxygenator including search for thrombotic material

CONTACTS AND LOCATIONS:
Overall Officials: Onnen Moerer, Prof., Principal Investigator — Department of Anesthesiology, University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided